CLINICAL TRIAL: NCT02809118
Title: Efficacy and Safety of AM-111 as Acute Sudden Sensorineural Hearing Loss Treatment
Acronym: ASSENT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Availability of relevant new efficacy data from another study
Sponsor: Auris Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-111-CL-15-01
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-06

CONDITIONS: Hearing Loss, Idiopathic Sudden Sensorineural
Keywords: Deafness; Hearing Loss; Hearing Loss, Sensorineural; Ear Diseases; Hearing Disorders; Nervous System Diseases; Neurologic Manifestations; Otorhinolaryngologic Diseases; Sensation Disorders; Signs and Symptoms; Hearing and Speech Impairment; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Loss, Sensorineural; Ear Diseases; Hearing Disorders; Nervous System Diseases; Neurologic Manifestations; Otorhinolaryngologic Diseases; Sensation Disorders; Signs and Symptoms; Speech Disorders; Hearing Loss, Unilateral | interventions — D-JNKI-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo gel for intratympanic use
  Interventions: Other: Placebo
- AM-111 0.4 mg/ml (Experimental): AM-111 gel for intratympanic use (0.4 mg/ml AM-111)
  Interventions: Drug: AM-111 0.4 mg/ml
- AM-111 0.8 mg/ml (Experimental): AM-111 gel for intratympanic use (0.8 mg/ml AM-111)
  Interventions: Drug: AM-111 0.8 mg/ml

INTERVENTIONS:
Drug: AM-111 0.4 mg/ml — AM-111 0.4 mg/mL gel is administered with a single dose into the affected ear after topical anesthesia
  Other Names: Brimapitide
  Arms: AM-111 0.4 mg/ml
Drug: AM-111 0.8 mg/ml — AM-111 0.8 mg/mL gel is administered with a single dose into the affected ear after topical anesthesia
  Other Names: Brimapitide
  Arms: AM-111 0.8 mg/ml
Other: Placebo — Placebo gel is administered with a single dose into the affected ear after topical anesthesia
  Arms: Placebo

SUMMARY:
The primary objective of the trial is the confirmation of the efficacy of AM-111 in the recovery of severe to profound idiopathic sudden sensorineural hearing loss (ISSNHL).

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, parallel group, multi-center, efficacy and safety trial of AM-111 in the treatment of subjects suffering from severe to profound idiopathic sudden sensorineural hearing loss.

The active pharmaceutical ingredient of AM-111 is a JNK inhibitor (D-JNKI-1), a synthetic peptide consisting of 31 D-amino acids, which acts as a c-Jun N-terminal kinase (JNK) ligand.

The study consists of one treatment visit and a follow-up period until day 91.

Study participants will receive, after topical anesthesia of the tympanic membrane, AM-111 0.4 mg/mL or 0.8 mg/mL or placebo, administered into the affected ear. Following the administration, subjects will rest in a supine or reclined position for 30 minutes. Study participants will have the option for a course of oral corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral idiopathic sudden sensorineural hearing loss (ISSNHL) with onset within 72 hours prior to study treatment;
2. Mean hearing threshold of equal to or worse than (≥) 60 dB averaged across those 3 contiguous air conduction audiometric pure tone frequencies that show the highest mean hearing loss compared with the unaffected contralateral ear or, in case of history of asymmetric hearing, corresponding values from a pre-existing audiogram for the affected ear not older than 2 years prior to the ISSNHL incident (defined as "pure tone average", PTA);
3. Mean hearing loss of equal to or worse than (≥) 40 dB averaged across the air conduction thresholds at the pure tone average frequencies compared with the unaffected contralateral ear or, in case of history of asymmetric hearing, corresponding values from a preexisting audiogram for the affected ear not older than 2 years prior to the ISSNHL incident;
4. Age ≥ 18 years on the day of screening;

Exclusion Criteria:

1. Bilateral ISSNHL;
2. Acute hearing loss from noise trauma, barotrauma or head trauma;
3. Air-bone gap greater than 20 dB at the average of 3 contiguous test frequencies below 4 kHz, when the air-bone gap is measurable;
4. History of autoimmune hearing loss, radiation-induced hearing loss, endolymphatic hydrops or Menière's disease in either ear;
5. History of chronic inflammatory or suppurative ear disease or cholesteatoma in the affected ear;
6. Current evidence or history of acoustic neuroma or other retrocochlear damage in the affected ear;
7. History of otosclerosis in the affected ear;
8. Suspected perilymph fistula or membrane rupture in the affected ear;
9. Congenital hearing loss;
10. History of ISSNHL in the past 2 years;
11. Otitis media or otitis externa that is ongoing or ended within 7 days prior to study treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meier, Study Director — Auris Medical, Inc.
Locations (46):
- United States (37):
  - Birmingham, Alabama
  - Escondido, California
  - Fresno, California
  - La Jolla, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Celebration, Florida
  - Miami, Florida
  - Port Saint Lucie, Florida
  - Chicago, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Novi, Michigan
  - Columbia, Missouri
  - Lebanon, New Hampshire
  - Charlotte, New York
  - New Hyde Park, New York
  - New Windsor, New York
  - New York, New York
  - Rochester, New York
  - White Plains, New York
  - Matthews, North Carolina
  - Winston-Salem, North Carolina
  - Havertown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Lugoff, South Carolina
  - Orangeburg, South Carolina
  - Nashville, Tennessee
  - Fort Sam Houston, Texas
  - Salt Lake City, Utah
  - St. George, Utah
  - Norfolk, Virginia
  - Tacoma, Washington
- Canada (3):
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Markham, Ontario
- South Korea (6):
  - Seongnam-si, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Incheon, Jung-Gu
  - Gwangju
  - Pusan
  - Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was prematurely discontinued while recruitment was still low (56 out of the planned 300 subjects).
  Recruitment started on 16 June 2016. On 28 November 2017, recruitment was stopped. This study was conducted in USA, Canada and South Korea.
Pre-assignment Details: In subjects assessed within the first 24 hours from Idiopathic Sudden Sensorineural Hearing Loss (ISSNHL) onset, mean hearing threshold had to be confirmed by a second measure that was conducted, at the earliest, 24 hours after the onset of ISSNHL.
Period: Overall Study
Arm/Group | Placebo | AM-111 0.4 mg/ml | AM-111 0.8 mg/ml
Started | 18 | 19 | 19
Completed | 18 | 18 | 18
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AM-111 0.4 mg/ml | AM-111 0.8 mg/ml | Total
Number analyzed (Participants) | 18 | 19 | 19 | 56
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 57.7 (15.25) | 57.0 (15.13) | 54.6 (14.36) | 55.6 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 8 | 27
  Male | 6 | 12 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 8 | 11 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 6 | 10 | 6 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pure Tone Average (PTA)
Description: Measurement of the recovery of hearing between Day 0 (before treatment) and Day 91, i.e. change in pure tone audiometry between Day 0 and Day 91. The study was prematurely terminated. It was pre-specified not to complete analyses due to premature termination. Not all data planned were collected. No meaningful efficacy analysis could be performed on the data.
Time Frame: Day 0 and Day 91: The study was prematurely terminated.
Population: The study was prematurely terminated. No meaningful efficacy analysis could be performed on the data.
Arm/Group | Placebo | AM-111 0.4 mg/ml | AM-111 0.8 mg/ml
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Word Recognition Score (WRS) - Main Secondary
Description: Change in WRS from Day 0 to Day 91. The WRS was determined with country-/language-specific word lists. At least 20 mono- or disyllabic words were presented in random order. After each word was presented to the subject, the subject was asked to repeat it, and to guess it, if he/she was not sure of the word. The study was prematurely terminated. It was pre-specified not to complete analyses due to premature termination. Not all data planned were collected. No meaningful efficacy analysis could be performed on the data.
Time Frame: Day 0 and Day 91: The study was prematurely terminated.
Population: The study was prematurely terminated. No meaningful efficacy analysis could be performed on the data.
Units Other Than Participants: Percentage of correct word responses
Arm/Group | Placebo | AM-111 0.4 mg/ml | AM-111 0.8 mg/ml
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (Percentage of correct word responses) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected from day 0 to day 91(±7).
Arm/Group | Placebo | AM-111 0.4 mg/ml | AM-111 0.8 mg/ml
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 8/18 | 11/19 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | AM-111 0.4 mg/ml (N=19) | AM-111 0.8 mg/ml (N=19)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | AM-111 0.4 mg/ml (N=19) | AM-111 0.8 mg/ml (N=19)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube disfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscoloskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mastocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic dilation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colour blindness (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspesia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02809118/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02809118/SAP_001.pdf